CLINICAL TRIAL: NCT07369635
Title: A Phase III, Multicenter, Randomized, Open-label, Parallel-controlled Clinical Trial Evaluating the Efficacy and Safety of Trĩ Thiên Dược Capsules in Grade II Internal Haemorrhoids Patients With Bleeding Compared to Diosmin.
Brief Title: A Phase III Clinical Trial Evaluating the Efficacy and Safety of TriThien Duoc Capsules in Grade II Internal Haemorrhoids Patients With Bleeding Compared to Diosmin.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 65/CN-HĐĐĐ
Record Dates: First submitted 2026-01-18; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-03

CONDITIONS: Grade II Internal Hemorrhoids With Bleeding
Keywords: Tri Thien Duoc; internal hemorrhoids; Portulaca Oleracea L.; Amaranthus Spinosus L.
MeSH Terms: interventions — Control Groups; Diosmin

STUDY DESIGN:
Intervention Model Description: A total of 172 participants with grade II internal hemorrhoids with bleeding were enrolled in the study and allocated as follows:
  Intervention Group: 86 participants received Tri Thien Duoc pills at a dosage of 8 capsules per day for 28 days, with follow-up conducted for 35 days from the initiation of treatment.
  Control Group: 86 participants received Diosmin (Daflon) at a dosage of 4 pills per day for 28 days, with follow-up conducted for 35 days from the initiation of treatment.
  All participants in this Phase III study adhered to the dietary and lifestyle recommendations outlined by the American Gastroenterological Association for hemorrhoid management, including:
  Maintaining a high-fiber diet rich in vegetables and soft foods. Ensuring adequate hydration (1.5-2 litres of water per day). Engaging in regular physical activity. Avoiding prolonged sitting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tri Thien Duoc capsules (Experimental): Intervention Group: 86 participants with stage II hemorrhoids with bleeding
  Interventions: Drug: Intervention Group: Tri Thien Duoc Capsules
- Diosmin (Active Comparator): Control group: 86 participants with stage II hemorrhoids with bleeding
  Interventions: Drug: Control group (diosmin)

INTERVENTIONS:
Drug: Intervention Group: Tri Thien Duoc Capsules — Intervention Group: 86 participants received Tri Thien Duoc pills at a dosage of 8 capsules per day for 28 days, with follow-up conducted for 35 days from the initiation of treatment.
  Arms: Tri Thien Duoc capsules
Drug: Control group (diosmin) — Control group: 86 patients took Daflon, 4 tablets/day for 28 days, monitored for 35 days from the start of treatment.
  Arms: Diosmin

SUMMARY:
A Phase III, randomized, double-blind, placebo-controlled clinical trial has been conducted to evaluate the efficacy and safety of Trĩ Thiên Dược capsules in people with grade II internal hemorrhoids with bleeding. This study aims to further assess the therapeutic effects and potential adverse effects of Trĩ Thiên Dược, a herbal formulation containing Portulaca Oleracea L. (purslane) and Amaranthus Spinosus L. (spiny amaranth), in comparison to Diosmin (Daflon).Participants will undergo a 5-week study period and will be randomly assigned (1:1 ratio) into one of two groups:Research Group: Participants receiving Trĩ Thiên Dược tablets.Control Group: Participants receiving Daflon (Diosmin).The treatment regimen will last for 28 days, followed by an additional follow-up period extending to day 35 after the initial treatment.

DETAILED DESCRIPTION:
Study Design:

This study is a randomized, open-label, placebo-controlled trial evaluating the efficacy of Diosmin (Daflon) in people with grade II internal hemorrhoids with bleeding. Participants are randomly assigned in a 1:1 ratio to receive either Tri Thien Duoc pills or Diosmin (Daflon).

Participants:

A total of 172 participants with grade II internal hemorrhoids with bleeding were enrolled in the study and allocated as follows:

Intervention Group: 86 participants received Tri Thien Duoc pills at a dosage of 8 capsules per day for 28 days, with follow-up conducted for 35 days from the initiation of treatment.

Control Group: 86 participants received Diosmin (Daflon) at a dosage of 4 pills per day for 28 days, with follow-up conducted for 35 days from the initiation of treatment.

Study Procedures:

All participants in this Phase III study adhered to the dietary and lifestyle recommendations outlined by the American Gastroenterological Association for hemorrhoid management, including:

Maintaining a high-fiber diet rich in vegetables and soft foods. Ensuring adequate hydration (1.5-2 litres of water per day). Engaging in regular physical activity. Avoiding prolonged sitting.

Assessments and Monitoring:

Participants underwent clinical evaluations and monitoring throughout the study. Key clinical parameters were assessed at four-time points:

Baseline (Day 0, D0) Mid-treatment (Day 14, D14) End of treatment (Day 28, D28) Post-treatment follow-up (Day 35, D35) Laboratory tests, including liver and kidney function assessments, complete blood count, urinalysis, and colonoscopy, were conducted at baseline (D0) and treatment's end (D28).

ELIGIBILITY:
- Inclusion Criteria

Patients must meet all of the following criteria to be eligible for the study:

* Age 18 to 65 years
* Diagnosis of grade II internal hemorrhoids with bleeding, presenting with the following symptoms:

Hemorrhoids prolapse with gentle straining and retract spontaneously Presence of blood in stool Congested and/or bleeding hemorrhoids

* Having symptoms such as anal pain and anal itching
* Willingness to voluntarily participate in the study - Exclusion Criteria

Patients meeting any of the following criteria will be excluded from the study:

* History of malignancy, including colon cancer and other cancers
* Anal polyps and proctitis
* Anal fissures with bleeding
* Systemic diseases, such as hypertension, liver failure, kidney failure, heart failure, and coagulation disorders.
* Other severe acute or chronic illnesses
* Mixed hemorrhoids or conditions requiring immediate surgical intervention, such as hematoma, severe bleeding, or hemorrhoidal infarction
* Recent use of other hemorrhoid medications (within 7 days prior to study enrollment)
* Known allergy to any component of the study medications
* Pregnant or lactating women
* Patients will be withdrawn from the study if they: Do not adhere to the treatment regimen, including missing medication for more than 3 consecutive days. Or Use other prohibited medications during the study period. Or require routine medical care at the hospital due to non-compliance or other medical reasons.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Mean duration of rectal bleeding | Baseline (Day 0, start of treatment) End of treatment (Day 28, after 28 days of treatment) Follow-up (Day 35, 7 days post-treatment)
  Mean duration of fresh rectal bleeding episodes: Defined as the mean number of days the patient experiences fresh rectal bleeding.
Rate of cessation of rectal bleeding | Baseline (Day 0, start of treatment) End of treatment (Day 28, after 28 days of treatment) Follow-up (Day 35, 7 days post-treatment)
  Defined as the proportion of patients who achieve complete cessation of fresh rectal bleeding out of the total number of patients
Severity of hemorrhoidal symptoms | Baseline (Day 0, start of treatment) End of treatment (Day 28, after 28 days of treatment) Follow-up (Day 35, 7 days post-treatment)
  the mean symptom score of participants according to the Sodergren scale.

SECONDARY OUTCOMES:
Pain score during defecation | Baseline (Day 0, start of treatment) End of treatment (Day 28, after 28 days of treatment) Follow-up (Day 35, 7 days post-treatment)
  The average pain level score reported by patients during defecation, measured using the Visual Analog Scale (VAS).
Rate of recurrent bleeding | During 35 days of follow up
  The number of patients experiencing rebleeding out of the total number of patients in each group.
Degree of defecation disorder | Baseline (Day 0, start of treatment) End of treatment (Day 28, after 28 days of treatment) Follow-up (Day 35, 7 days post-treatment)
  The average Wexner Defecation Disorder Score, which quantifies the severity of defecation dysfunction.
Degree of hemorrhoid prolapse | Baseline (Day 0, start of treatment); End of treatment (Day 28, after 28 days of treatment)
  the proportion of patients classified according to each degree of hemorrhoid severity, as determined by clinical examination and rigid sigmoidoscopy.
Anal mucosal condition | Baseline (Day 0, start of treatment); End of treatment (Day 28, after 28 days of treatment)
  The percentage of patients classified according to the degree of hemorrhoidal engorgement, as assessed by rigid sigmoidoscopy.
Adverse Events | During 28 days of treatment
  the proportion of patients who experienced a drug-related adverse event during the study period in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
All IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 3 years after the publication of results
Access Criteria: * Criteria for Data Sharing:
    * Data will only be shared if it serves a valid scientific purpose (e.g., verifying results, conducting meaningful new analyses).
    * The statistical methods must be reviewed and approved by experts or an independent committee before use.
  * Mechanism for Data Sharing:
    * Researchers must submit a proposal describing their study and analysis methods.
    * They must sign a confidentiality and data use agreement.
    * Once approved, the data will be provided through a secure system